## APPROVED BY THE YALE UNIVERSITY IRB 1/8/2021

## HIC 2000028482; NCT04630054

## Face Masks to Reduce COVID-19 in Bangladesh Study Consent Script

As-salamua-likum, sir. My name is \${enumname}. I am working for Innovations for Poverty Action (IPA) - a non-profit organization. In collaboration with Bangladesh Government's Access to Information (IPA), Informed Consent Script for Participation in Research Study research to understand how (this will be used during iscarciting study participants from resident in this community, we would like to invite you to participate in this study.

## communities)

If you agree to participate in this study, we will ask for your contact information so we can interview you several times in the next 4 months. During these interviews, we will ask you questions about your health and thins you do to reduce your health risk for 10-15 minutes. Your answers will be anonymously combined with the answers of other people in your community and people from many other communities. We will use the responses to inform organizations such as the government, BRAC, and healthcare providers how to best protect you and your community.

As part of the study, we will also determine whether some participants have been exposed to coronavirus and other diseases. If you are selected to be tested, we will give you more details later on and will ask for your further consent before proceeding with any tests.

Participation is voluntary and you can withdraw your participation anytime or refuse to answer any question or stop the interview at any time. Refusal to participate will not result in any penalty or loss of existing benefits.

All your responses will be confidential and protected. Your answers will never be shared with your neighbors or the community. Information that identifies you will not be shared outside of research teams from IPA and Yale.

Your information will not be used for future research studies or distributed to another investigator for future research studies without additional informed consent from you.

As researchers, we cannot provide you any direct benefit. This is a research study so we do not provide healthcare. However, your participation will help us learn how the spread of infectious diseases can be reduced and that learning might help the government and NGOs to fight the current and future pandemics.

Do you have any questions about the study?

If you have a question later, or if you have concerns or complaints about this interview, please contact Mr. Alamgir Kabir, Senior Operations Manager, Innovations for Poverty Action, Phone +8801712121221 or Mr. Mohammad Ashraful Haque, Bangladesh Country Director, Innovations for Poverty Action, Phone +8801913973321. You can also share your concerns or complaints with the Bangladesh Medical Research Council by contacting info@bmrcbd.org.

Are you willing to participate in the study?